CLINICAL TRIAL: NCT00633217
Title: A Randomized, Double-Blind, Double-Dummy, Parallel Group 12-Week Comparison of the Efficacy and Safety of Fluticasone Propionate/Salmeterol Hydrofluoroalkane 134a Metered-Dose-Inhaler 230/42mcg Twice-daily With Fluticasone Propionate/Salmeterol DISKUS 250/50mcg Twice-daily in Subjects With COPD
Brief Title: Advair HFA For Chronic Obstructive Pulmonary Disease(COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111117
Record Dates: First submitted 2008-02-19; First posted 2008-03-11 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: DISKUS; Salmeterol; Fluticasone Propionate; Chronic Obstructive Pulmonary Disease (COPD); Hydroflouroalkane; COPD; HFA MDI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- arm 1 (Active Comparator)
  Interventions: Drug: Fluticasone Propionate/Salmeterol DISKUS 250/50mcg
- arm 2 (Experimental)
  Interventions: Drug: Fluticasone Propionate/Salmeterol Hydrofluoroalkane 134a MDI 230/42mcg

INTERVENTIONS:
Drug: Fluticasone Propionate/Salmeterol DISKUS 250/50mcg — treatment drug
  Arms: arm 1
Drug: Fluticasone Propionate/Salmeterol Hydrofluoroalkane 134a MDI 230/42mcg — treatment drug
  Other Names: Fluticasone Propionate/Salmeterol DISKUS 250/50mcg
  Arms: arm 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the FSC HFA MDI in subjects with COPD. The dose of FSC HFA MDI to be evaluated corresponds to the dose of FSC DISKUS (250/50mcg twice-daily) that is indicated for the treatment of COPD associated with chronic bronchitis in the US. This study will last up to approximately 15 weeks, and subjects will visit the clinic 5 times. Subjects will be given breathing tests and will record their peak expiratory flow measurements daily on diary cards. All study related medicines and medical examinations will be provided at no cost. The FSC HFA MDI used in this study has been approved by FDA for use in asthma while the FSC 250/50mcg DISKUS has been approved for use in asthma and COPD.

ELIGIBILITY:
Inclusion criteria:

Subjects eligible for enrollment in the study must meet all of the following criteria:

* Signed and dated written informed consent obtained from the subject and/or subject's legally acceptable representative prior to study participation.
* Males or females ≥ 40 years of age.

A female is eligible to participate in this study if she is of:

1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal [i.e., >1 year without menses in the absence of hormone replacement therapy]); or,
2. child-bearing potential, has a negative pregnancy test (urine) at screen, and one of the following applies:

   * Abstinence from intercourse, or,
   * Male partner was sterile prior to the female subject's entry into the study, or,
   * Use of implants of levonorgestrel; or,
   * Injectable progesterone; or,
   * Oral contraceptive (combined or progesterone only), contraceptive patch, vaginal ring; or,
   * Any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year (e.g., Paragard), or,
   * Double barrier technique simultaneously using two of the following: spermicide, male condom, diaphragm, or female condom

     * An established clinical history of COPD (including chronic bronchitis and/or emphysema) in accordance with the following definition by the American Thoracic Society:

COPD is a preventable and treatable disease state characterised by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences [Celli, 2004].

* A post-albuterol FEV1/FVC ratio of ≤ 0.70
* A post-albuterol FEV1 ≥ 0.70L and ≤ 70% of predicted normal OR a post-albuterol FEV1 of ≤ 0.70L and ≥40% of predicted normal but still ≤70% of predicted normal based on NHANES III reference values [Hankinson, 1999].
* Current or previous smokers with a cigarette smoking history of ≥ 10 pack-years. [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 10 pack-years is equal to 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years]. Former-smokers are defined as subjects who have discontinued smoking for ≥ 6 months prior to Visit 1. Subjects who decide to stop smoking at Visit 1 will not be eligible for participation in the study.

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* A current diagnosis of asthma.
* Any clinically significant and uncontrolled disease, including but not limited to the following: neurological, psychiatric, renal, immunological, endocrine/metabolic (including uncontrolled diabetes, hypokalemia or thyroid disease), cardiovascular, neuromuscular, hepatic, gastric, or hematological abnormalities, or peripheral vascular disease. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would affect the efficacy analysis if the disease/condition exacerbated during the study.
* A respiratory diagnosis other than COPD (e.g., lung cancer, bronchiectasis, sarcoidosis, tuberculosis, lung fibrosis), including subjects with a diagnosis of alpha-1-antitrypsin deficiency. Allergic rhinitis is not exclusionary.
* An abnormal and clinically significant chest x-ray or computed tomography (CT) scan not believed to be due to the presence of COPD. A chest x-ray must be taken if the subject has not had one within 6 months of Visit 1.
* An abnormal and clinically significant 12-lead electrocardiogram (ECG). For the purposes of this study, an abnormal ECG is defined as a 12-lead tracing which is interpreted with (but not limited to) any of the following:

  * Myocardial ischemia
  * Clinically significant conduction abnormalities (e.g., left bundle branch block, Wolff-Parkinson-White syndrome)
  * Clinically significant arrhythmias (e.g., atrial fibrillation, ventricular tachycardia) The study investigator will determine the clinical significance of any ECG abnormality and determine if a subject is precluded from entering the study.
* Previously diagnosed cancer unless it is in complete clinical remission (no evidence of any tumor burden) at Visit 1. Localized carcinomas of the skin that have been resected for cure are not considered exclusionary.
* Any immediate or delayed hypersensitivity to any beta-agonist, sympathomimetic drug, or intranasal, inhaled, or oral corticosteroid including any components of the formulations (e.g. lactose or milk protein).
* Initiation of systemic beta-blocker medications within 30 days of Visit 1.
* Use of products containing the protease inhibitor ritonavir (Norvir, Kaletra).
* Use of the following medications within the defined times prior to Visit 1:

Medication (Exclusion Prior to Visit 1) Short-acting beta-agonists (e.g., albuterol) (6 hours) Ipratropium (6 hours) Ipratropium/albuterol combination product (6 hours) Oral beta-agonists (48 hours) Salmeterol and formoterol (48 hours) Theophylline preparations (48 hours) Tiotropium (48 hours) Long-acting beta-agonist/inhaled corticosteroid combination products (e.g., ADVAIR™ or Symbicort) (30 days) Inhaled corticosteroids (30 days) Oral or parenteral corticosteroids (30 days) Any investigational drug (30 days)

* Lung resection surgery (e.g., lung volume reduction surgery, or lobectomy) within 1 year of Visit 1.
* A COPD exacerbation and/or infection of the upper or lower respiratory tract requiring treatment with systemic (oral or parenteral) corticosteroids and/or antibiotics that has not resolved within 30 days of Visit 1
* A COPD exacerbation that resulted in hospitalization that has not resolved within 3 months of Visit 1.
* Use of nocturnal positive pressure [e.g., continuous positive airway pressure or bi-level positive airway pressure].
* A body mass index (BMI) of ≥ 40kg/m².
* Subject is a study investigator, sub-investigator, study coordinator, or employee of a participating investigator or immediate family members of the aforementioned.
* Any intellectual deficiency including illiteracy, history of substance abuse in the two years prior to Visit 1 (including drug and alcohol), or other conditions, which will limit the validity of informed consent to participate in the study.
* Supplemental oxygen, with the following exceptions:

  * Use at high altitude (> 5000 feet) provided subject does not require a flow rate of > 2 L/minute
  * Use for exertion provided subject does not require > 2 hours per day of oxygen and does not require a flow rate of > 2L/minute
  * Use for nocturnal therapy provided subject does not require a flow rate of > 2L/minute

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (16):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Koser A, Westerman J, Sharma S, Emmett A, Crater GD. Safety and efficacy of fluticasone propionate/salmeterol hydrofluoroalkane 134a metered-dose-inhaler compared with fluticasone propionate/salmeterol diskus in patients with chronic obstructive pulmonary disease. Open Respir Med J. 2010 Oct 21;4:86-91. doi: 10.2174/1874306401004010086. PMID 21253451
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- HFA MDI 230/42 mcg and Matching DISKUS Placebo: Fluticasone Propionate/Salmeterol Hydrofluoroalkane (HFA) 134a metered-dose inhaler (MDI) 230/42 micrograms (mcg) twice daily and matching DISKUS placebo
- DISKUS 250/50 mcg and Matching HFA MDI Placebo: Fluticasone Propionate/Salmeterol DISKUS 250/50 mcg twice daily and matching HFA MDI placebo
Period: Overall Study
Arm/Group | HFA MDI 230/42 mcg and Matching DISKUS Placebo | DISKUS 250/50 mcg and Matching HFA MDI Placebo
Started | 121 | 126
Completed | 106 | 103
Not Completed | 15 | 23
Not completed — Adverse Event | 5 | 9
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 3 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Investigator Discretion | 2 | 0
Not completed — Withdrew Consent | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HFA MDI 230/42 mcg and Matching DISKUS Placebo | DISKUS 250/50 mcg and Matching HFA MDI Placebo | Total
Number analyzed (Participants) | 121 | 126 | 247
Age, Continuous [Mean (Full Range); unit: years] | 61.6 [40 to 84] | 63.4 [45 to 86] | 61.6 [40 to 86]
Gender [Count of Participants; unit: Participants]
  Female | 55 | 60 | 115
  Male | 66 | 66 | 132
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 10 | 9 | 19
  White - White/Caucasian/European Heritage | 109 | 117 | 226
  American Indian or Alaskan Native | 1 | 0 | 1
  White - Arabic/North African Heritage | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Forced Expiratory Volume in One Second (FEV1) 2 Hours Post-dose of Blinded Study Drug
Description: The primary efficacy analysis was mean change from baseline in 2-hour post-dose FEV1 compared between the two treatment groups at Endpoint. Change from baseline was calculated as the value at Endpoint minus the baseline value. FEV1, which is assessed using spirometry, is the maximal amount of air you can forcefully exhale in one second. Endpoint was defined as the last scheduled observation for 2 hour post-dose FEV1 during the 12-week treatment period.
Time Frame: 2 hours after administration of blinded study drug; Baseline through Week 12
Population: Intent-to-Treat (ITT) Population: all participants who had been randomized to study drug. The numbers analyzed do not match Baseline numbers due to missing data for some participants.
Measure: Mean (Standard Error); unit: milliliters (mL)
Arm/Group | HFA MDI 230/42 mcg and Matching DISKUS Placebo | DISKUS 250/50 mcg and Matching HFA MDI Placebo
Number analyzed (Participants) | 116 | 115
milliliters (mL) | 155 (23.4) | 150 (21.9)
Statistical Analysis 1: Comparison: HFA MDI 230/42 mcg and Matching DISKUS Placebo vs DISKUS 250/50 mcg and Matching HFA MDI Placebo; Test type: Non-Inferiority or Equivalence — If the lower bound of the 95% confidence interval for the mean difference in 2-hour post-dose FEV1 change from baseline fell above -75 mL, then HFA MDI could be deemed non-inferior to DISKUS treatment response; p = 0.021, ANCOVA

2. Secondary Outcome: Mean Change From Baseline in AM Pre-dose FEV1
Description: Change from baseline was calculated as the value at Endpoint minus the baseline value. AM pre-dose FEV1, which is assessed using spirometry, is the maximum amount of air you can forcefully exhale in one second prior to taking the morning dose of study drug. Endpoint was defined as the last scheduled observation for AM pre-dose FEV1 during the 12-week treatment period.
Time Frame: Measurement of FEV1 prior to study drug administration; Baseline through Week 12
Population: ITT Population. The numbers analyzed do not match Baseline numbers due to missing data for some participants.
Measure: Mean (Standard Error); unit: mL
Arm/Group | HFA MDI 230/42 mcg and Matching DISKUS Placebo | DISKUS 250/50 mcg and Matching HFA MDI Placebo
Number analyzed (Participants) | 116 | 115
mL | 74 (20.6) | 77 (20.5)

3. Secondary Outcome: Mean Change From Baseline in Peak Expiratory Flow
Description: The peak expiratory flow is a measure of the amount of air that can be pushed through the airways in a single rapid exhalation. This is measured by a peak flow meter which is a hand held device. Change from baseline was calculated as the average value over Weeks 1-12 minus the baseline value.
Time Frame: Baseline through Week 12
Population: ITT Population. Some participants did not have measured values for peak expiratory flow and were thus not included in the analysis.
Measure: Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | HFA MDI 230/42 mcg and Matching DISKUS Placebo | DISKUS 250/50 mcg and Matching HFA MDI Placebo
Number analyzed (Participants) | 119 | 116
Liters/minute (L/min) | 21.8 (2.66) | 18.7 (2.48)

ADVERSE EVENTS:
Arm/Group | HFA MDI 230/42 mcg and Matching DISKUS Placebo | DISKUS 250/50 mcg and Matching HFA MDI Placebo
Serious Adverse Events (participants affected / at risk) | 6/121 | 3/126
Other Adverse Events (participants affected / at risk) | 27/121 | 29/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HFA MDI 230/42 mcg and Matching DISKUS Placebo (N=121) | DISKUS 250/50 mcg and Matching HFA MDI Placebo (N=126)
Chronic Obstructive Pulmonary Disease Exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HFA MDI 230/42 mcg and Matching DISKUS Placebo (N=121) | DISKUS 250/50 mcg and Matching HFA MDI Placebo (N=126)
Headache (Nervous system disorders) | 10 | 8
Nasopharyngitis (Infections and infestations) | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Sinusitis (Infections and infestations) | 3 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.